CLINICAL TRIAL: NCT01712906
Title: A Phase II Clinical Trial for Live Attenuated Mumps (F-genotype) Vaccine (Human Diploid Cell, KMB-17) in Chinese Children
Brief Title: A Phase I, Safety Study of Live Attenuated Mumps (F-genotype) Vaccine (Human Diploid Cell, KMB-17) in Chinese Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Institute of Medical Biology, Chinese Academy of Medical Sciences (Other)
Collaborators: Hebei Provincial Center for Diseases Control and Prevention (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: FMumps-KMB17-I-IMB-CAMS
Record Dates: First submitted 2012-10-22; First posted 2012-10-24 (Estimated); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Mumps
Keywords: Live Attenuated Mumps (F-genotype) Vaccine
MeSH Terms: conditions — Mumps | interventions — Long-Term Synaptic Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (18):
- 3.50±0.25logCCID50/ml in adults (Experimental): Attenuated Mumps vaccine (KMB-17) of 3.50±0.25logCCID50/ml in 16 adults aged 16-59 years old on day 0.
  Interventions: Biological: 3.50±0.25logCCID50/ml
- 4.25±0.25 logCCID50/ml in adults (Experimental): Attenuated Mumps vaccine (KMB-17) of 4.25±0.25 logCCID50/ml in 16 adults aged 16-59 years old on day 0.
  Interventions: Biological: 4.25±0.25 logCCID50/ml
- 5.00±0.25 logCCID50/ml in adults (Experimental): Attenuated Mumps vaccine (KMB-17) of 4.25±0.25 logCCID50/ml in 16 adults aged 16-59 years old on day 0.
  Interventions: Biological: 5.00±0.25 logCCID50/ml
- 0 logCCID50/ml in adults (Placebo Comparator): 0 logCCID50/ml in 18 adults aged 16-59 years old on day 0.
  Interventions: Biological: 0 logCCID50/ml
- 3.50±0.25logCCID50/ml in children (5-15 years old) (Experimental): Attenuated Mumps vaccine (KMB-17) of 3.50±0.25logCCID50/ml in 16 children aged 5-15 years old on day 0.
  Interventions: Biological: 3.50±0.25logCCID50/ml
- 4.25±0.25 logCCID50/ml in children (5-15 years old) (Experimental): Attenuated Mumps vaccine (KMB-17) of 4.25±0.25 logCCID50/ml in 16 children aged 5-15 years old on day 0.
  Interventions: Biological: 4.25±0.25 logCCID50/ml
- 5.00±0.25 logCCID50/ml in children (5-15 years old) (Experimental): Attenuated Mumps vaccine (KMB-17) of 5.00±0.25 logCCID50/ml in 16 children aged 5-15 years old on day 0.
  Interventions: Biological: 5.00±0.25 logCCID50/ml
- 0 logCCID50/ml in children (5-15 years old) (Placebo Comparator): 0 logCCID50/ml in 18 children aged 5-15 years old on day 0.
  Interventions: Biological: 0 logCCID50/ml
- 3.50±0.25logCCID50/ml in children (2-4 years old) (Experimental): Attenuated Mumps vaccine (KMB-17) of 3.50±0.25logCCID50/ml in 16 children aged 2-4 years old on day 0.
  Interventions: Biological: 3.50±0.25logCCID50/ml
- 4.25±0.25 logCCID50/ml in children (2-4 years old) (Experimental): Attenuated Mumps vaccine (KMB-17) of 4.25±0.25 logCCID50/ml in 16 children aged 2-4 years old on day 0.
  Interventions: Biological: 4.25±0.25 logCCID50/ml
- 5.00±0.25 logCCID50/ml in children (2-4 years old) (Experimental): Attenuated Mumps vaccine (KMB-17) of 5.00±0.25 logCCID50/ml in 16 children aged 2-4 years old on day 0.
  Interventions: Biological: 5.00±0.25 logCCID50/ml
- 0 logCCID50/ml in children (2-4 years old) (Placebo Comparator): 0 logCCID50/ml in 18 children aged 2-4 years old on day 0.
  Interventions: Biological: 0 logCCID50/ml
- Attenuated Mumps vaccine in children (2-4 years old) (Active Comparator): Attenuated Mumps vaccine (Zhe Jiang Vacn Bio-pharmaceutical Co., LTD.; NO.20110528-1) in 18 children aged 2-4 years old on day 0.
  Interventions: Biological: Attenuated Mumps vaccine (Zhe Jiang Vacn Bio-pharmaceutical Co., LTD.; NO.20110528-1)
- 3.50±0.25logCCID50/ml in infants (Experimental): Attenuated Mumps vaccine (KMB-17) of 3.50±0.25logCCID50/ml in 16 infants aged 8-23 months old on day 0.
  Interventions: Biological: 3.50±0.25logCCID50/ml
- 4.25±0.25 logCCID50/ml in infants (Experimental): Attenuated Mumps vaccine (KMB-17) of 4.25±0.25 logCCID50/ml in 16 infants aged 8-23 months old on day 0.
  Interventions: Biological: 4.25±0.25 logCCID50/ml
- 5.00±0.25 logCCID50/ml in infants (Experimental): Attenuated Mumps vaccine (KMB-17) of 5.00±0.25 logCCID50/ml in 16 infants aged 8-23 months old on day 0.
  Interventions: Biological: 5.00±0.25 logCCID50/ml
- 0 logCCID50/ml in infants (Placebo Comparator): 0 logCCID50/ml in 18 infants aged 8-23 months old on day 0.
  Interventions: Biological: 0 logCCID50/ml
- Attenuated Mumps vaccine in infants (Active Comparator): Attenuated Mumps vaccine (Zhe Jiang Vacn Bio-pharmaceutical Co., LTD.; NO.20110528-1) in 18 infants aged 8-23 months old on day 0.
  Interventions: Biological: Attenuated Mumps vaccine (Zhe Jiang Vacn Bio-pharmaceutical Co., LTD.; NO.20110528-1)

INTERVENTIONS:
Biological: 3.50±0.25logCCID50/ml — Attenuated Mumps vaccine (KMB-17) of 3.50±0.25logCCID50/ml in adults (16-59 years old)，children (5-15 years old or 2-4 years old) and infants (8-23 months old) on day 0.
  Arms: 3.50±0.25logCCID50/ml in adults; 3.50±0.25logCCID50/ml in children (2-4 years old); 3.50±0.25logCCID50/ml in children (5-15 years old); 3.50±0.25logCCID50/ml in infants
Biological: 4.25±0.25 logCCID50/ml — Attenuated Mumps vaccine (KMB-17) of 4.25±0.25 logCCID50/ml in adults (16-59 years old)，children (5-15 years old or 2-4 years old) and infants (8-23 months old) on day 0.
  Arms: 4.25±0.25 logCCID50/ml in adults; 4.25±0.25 logCCID50/ml in children (2-4 years old); 4.25±0.25 logCCID50/ml in children (5-15 years old); 4.25±0.25 logCCID50/ml in infants
Biological: 5.00±0.25 logCCID50/ml — Attenuated Mumps vaccine (KMB-17) of 5.00±0.25 logCCID50/ml in adults (16-59 years old)，children (5-15 years old or 2-4 years old) and infants (8-23 months old) on day 0.
  Arms: 5.00±0.25 logCCID50/ml in adults; 5.00±0.25 logCCID50/ml in children (2-4 years old); 5.00±0.25 logCCID50/ml in children (5-15 years old); 5.00±0.25 logCCID50/ml in infants
Biological: 0 logCCID50/ml — 0 logCCID50/ml in adults (16-59 years old)，children (5-15 years old or 2-4 years old) and infants (8-23 months old) on day 0.
  Arms: 0 logCCID50/ml in adults; 0 logCCID50/ml in children (2-4 years old); 0 logCCID50/ml in children (5-15 years old); 0 logCCID50/ml in infants
Biological: Attenuated Mumps vaccine (Zhe Jiang Vacn Bio-pharmaceutical Co., LTD.; NO.20110528-1) — Attenuated Mumps vaccine (Zhe Jiang Vacn Bio-pharmaceutical Co., LTD.; NO.20110528-1) in children (2-4 years old) and infants (8-23 months old) on day 0.
  Arms: Attenuated Mumps vaccine in children (2-4 years old); Attenuated Mumps vaccine in infants

SUMMARY:
Mumps is an acute infectious respiratory disease caused by the mumps virus (MuV), which occurs mainly in children and adolescents. Its main clinical symptoms were parotid gland suppurative swelling and pain with fever. The pathological changes and harm caused by mumps was not only confined to the parotid gland, on the contrary, the social harm caused by serious complications cannot be ignored. As mumps is a vaccine-preventable infectious disease, vaccination is a fundamental strategy for controlling mumps. So far, there are 13 genotypes of MuV. Based on the analysis of molecular epidemiology, the main epidemic strain of MuV in China was the F genotype. The commonly used vaccine strains represented only a small number of known genotypes, e.g. Jeryl-Lynn (JL) and Rubini strains, which belong to type A, Urabe strain belongs to type B, and L-Zagreb strains belongs to type D. Virus seed of Live Attenuated Mumps Vaccine (Human diploid cell) developed by the institute was SP-A strain, which was the first separation and preparation of the attenuated mumps viruses in China. SP-A belongs to F genotype, which was the domestic epidemic genotype. In addition, the cell substrate prepared for vaccine was human diploid cell (KMB-17 strain), which is much safer to use. The preliminary test results showed that the vaccine possessed good immunogenicity and good antigenic cross-reactivity. The application of this vaccine will provide more effective means to prevent and control of mumps epidemic.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects (8 months-59 years old) as established by medical history and clinical examination
* The subjects oneself or their legal guardian must be aware of this vaccines
* Voluntarily participate in the study and signed Informed Consent Form
* Subjects with temperature ≤ 37.0℃
* With the ability and objective to comply with the requirements of the protocol
* Persist for a 1-month visit and receive blood tests according to program requirements

Exclusion Criteria:

* Subject who has a clinical diagnosis Mumps
* Subject who vaccinated Mumps vaccine in last 6 months
* ≤37 weeks gestation
* weight ≤ 2500 g when it was born
* Allergy or serious side-effects to a vaccine or any ingredient of vaccine
* Epilepsy, seizures, convulsions, neurological illness
* Congenital or hereditary immunodeficiency
* Autoimmune disease
* Severe malnutrition or dysgenopathy
* Asthma, thyroidectomy, angioneurotic edema, diabetes or cancer
* Asplenia, functional asplenia, and any circumstances leading to the asplenia or splenectomy
* Clinical diagnosis of coagulopathy (such as clotting factor deficiency, coagulation disorders, platelet abnormalities), significant bruising or blood clotting disorder
* Acute illness or acute exacerbation of chronic disease in last 7 days
* Any prior administration of immunodepressant or corticosteroids in last 6 months
* Any prior administration of blood products in last 3 months
* Any prior administration of live-attenuated vaccine in last 28 days or 1 months
* Any prior administration of subunit or inactivated vaccines in last 14 days
* Under the anti-TB prevention or therapy
* Fever before vaccination, axillary temperature ﹥37.0℃
* The laboratory test abnormalities before vaccination, including blood tests (hemoglobin, total white blood cells, WBC, platelets), blood biochemistry tests (ALT, total bilirubin, direct bilirubin, Cr, BUN) and urine tests (urine protein, urine sugar, blood cells), etc.
* Hypertension or hypotension. Systolic blood pressure ﹥140mmHg and/or diastolic blood pressure ﹥90mmHg; systolic blood pressure ﹤90mmHg and/or diastolic blood pressure ﹤60mmHg
* Breast-feeding, pregnant, planning a pregnancy within 60 days or positive pregnancy test women
* Any condition that in the opinion of the investigator, may interfere with the evaluation of study objectives

Ages: 8 Months to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 300 (Actual)
Dates: Start 2012-10; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Evaluate the Safety of Attenuated Mumps Vaccine (Human Diploid Cell, KMB-17) in Chinese Adults. | within the first 28 days after the vaccination
  Adverse reactions associated with vaccine were observed in Chinese Adults (from 16 to 59 years old) after the vaccination
Evaluate the Safety of Attenuated Mumps Vaccine (Human Diploid Cell, KMB-17) in Chinese Children. | within the first 28 days after the vaccination
  Adverse reactions associated with vaccine were observed in Chinese Children (from 5 to 15 years old) after the vaccination.
Evaluate the safety of Attenuated Mumps Vaccine (Human Diploid Cell, KMB-17) in Chinese Children. | within the first 28 days after the vaccination
  Adverse reactions associated with vaccine were observed in Chinese Children (from 2 to 4 years old) after the vaccination.
Evaluate the safety of Attenuated Mumps Vaccine (Human Diploid Cell, KMB-17) in Chinese Infants. | within the first 28 days after the vaccination
  Adverse reactions associated with vaccine were observed in Chinese Infants (from 8 to 23 months old) after the vaccination.

SECONDARY OUTCOMES:
Evaluate the seroconversion rate of anti-Mumps antibodies in serum of adults, children and infants, after vaccination. | within the first 28 days after the vaccination
  The seroconversion rate of anti-MuV antibodies was evaluated in serum of adults at the 0 and 28 days after vaccination.
  The seroconversion rate of anti-MuV antibodies was evaluated in serum of children at the 0 and 28 days after vaccination.
  The seroconversion rate of anti-MuV antibodies was evaluated in serum of infants at the 0 and 28 days after vaccination.
Evaluate the abnormity change of live and kidney function indexes in serum of adults, children and infants, after vaccination | within the first 4 days after the vaccination
  The abnormity change of live and kidney function indexes were evaluated in serum of adults at 0, 4 days after vaccination.
  The abnormity change of live and kidney function indexes were evaluated in serum of children at 0, 4 days after vaccination.
  The abnormity change of live and kidney function indexes were evaluated in serum of infants at 0, 4 days after vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Yuliang Zhao, Master, Principal Investigator — Hebei Provincial Center for Diseases Control and Prevention
Locations (1):
- Hebei Provincial Center for Diseases Control and Prevention, Shijiazhuang, Hebei, China

REFERENCES:
- [Derived] Liang Y, Ma J, Li C, Chen Y, Liu L, Liao Y, Zhang Y, Jiang L, Wang XY, Che Y, Deng W, Li H, Cui X, Ma N, Ding D, Xie Z, Cui P, Ji Q, Wang J, Zhao Y, Wang J, Li Q. Safety and immunogenicity of a live attenuated mumps vaccine: a phase I clinical trial. Hum Vaccin Immunother. 2014;10(5):1382-90. doi: 10.4161/hv.28334. Epub 2014 Mar 10. PMID 24614759